CLINICAL TRIAL: NCT01517620
Title: Total Glucosides Paeony Capsules in Maintaining Clinical Remission in Patients With Ankylosing Spondylitis Which Achieve Clinical Remission After Anti-TNF Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gu Jieruo, Department of Rheumatology, Third Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2011]2-38
Record Dates: First submitted 2012-01-15; First posted 2012-01-25 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total Glucosides Paeony, Capsules (Experimental)
  Interventions: Drug: Total Glucosides Paeony Capsules
- no intervention (No Intervention)

INTERVENTIONS:
Drug: Total Glucosides Paeony Capsules — Total Glucosides Paeony Capsules, oral, 0.3 gram per capsule, 3 capsules tid, 24 weeks
  Arms: Total Glucosides Paeony, Capsules

SUMMARY:
This is a prospective, randomized, open-label clinical trial to evaluate the efficacy and safety of total glucosides paeony capsules in maintaining clinical remission in patients with ankylosing spondylitis which achieved clinical remission after anti-TNF therapy. Patients will be divided into two groups randomly, one group receive non-steroid anti-inflammatory drugs(NSAID) mono-therapy and the other group receive total glucosides paeony capsules plus NSAID therapy for 24 weeks. The primary clinical endpoint is the proportion of patients which disease activity reaches relapse criteria. The investigator's hypothesis the proportion of relapse in total glucosides paeony capsules plus NSAID group would be lower than the NSAID mono-therapy group.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 16-65 years, sign the Informed Consent
* Fulfill 1984 modified NewYork classification criteria for AS
* Achieved clinical remission after at least 12 weeks' therapy of anti-TNF therapy
* Hb≥9g/dl, ALT/AST≤ 2 folds of upper level normal range, creatine≤120mol/L(≤1.4mg/dl)
* Commitment to contraceptive for woman

Exclusion Criteria:

* History of psoriasis and/or inflammatory bowel diseases
* Receive intra-articular injection of cortisone within 3 months before enrollment
* History of the listed diseases: heart failure, Multiple sclerosis, severe chronic obstructive pulmonary disease, frequent infections, lymphoma or other cancers, tuberculosis
* Pregnant and lactating women
* Mentally ill, Alcoholics and drug addicts

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
the proportion of patients which disease activity reaches relapse criteria | 24 weeks

SECONDARY OUTCOMES:
BASDAI score comparing to baseline | 24 weeks
BASFI score comparing to baseline | 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Rheumatology Department, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Rheumatology Department, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou